CLINICAL TRIAL: NCT06151119
Title: A Study to Evaluate 68Ga-FAPI PET/CT Imaging for Diagnosis, Grading, and Efficacy Evaluation of Myelofibrosis.
Brief Title: 68Ga-FAPI PET/CT Imaging for Diagnosis, Grading, and Efficacy Evaluation of Myelofibrosis.
Status: Recruiting | Type: Observational
Sponsor: The First Affiliated Hospital of Xiamen University (Other)
Responsible Party: Principal Investigator, Bing, Xu, Principal Investigator, The First Affiliated Hospital of Xiamen University
Other Study IDs: XMDYYYXYK-06
Record Dates: First submitted 2023-11-21; First posted 2023-11-30 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Primary Myelofibrosis
Keywords: Myelofibrosis; positron emission tomography / computed tomography
MeSH Terms: conditions — Primary Myelofibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- suspected or confirmed myelofibrosis: Patients with suspected or confirmed myelofibrosis;
  Interventions: Diagnostic Test: 68Ga FAPI PET/CT
- primary/secondary myelofibrosis: Patients with primary/secondary myelofibrosis who were not treated with ruxolitinib.
  Interventions: Diagnostic Test: 68Ga FAPI PET/CT

INTERVENTIONS:
Diagnostic Test: 68Ga FAPI PET/CT — 68Ga FAPI PET/CT

SUMMARY:
To evaluate the diagnostic efficacy of 68Ga FAPI PET/CT in myelofibrosis and to identify fibrosis grades.

To evaluate the diagnostic efficacy of 68Ga FAPIPET/CT imaging in patients with myelofibrosis, compared with conventional CT.

DETAILED DESCRIPTION:
This study uses bone marrow biopsy as a gold standard or reference standard to evaluate the diagnostic efficacy (Sensitivity, Specificity, Positive prediction rate, Negative prediction rate) of 68Ga FAPI PET/CT in myelofibrosis and to identify fibrosis grades.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old;
2. Cohort 1: Patients with suspected or confirmed myelofibrosis; Cohort 2: Patients with primary/secondary myelofibrosis who were not treated with ruxolitinib.
3. The expected survival time is over 3 months
4. Voluntarily sign informed consent.
5. Willing and able to follow the research protocol;
6. The subject must be able to lie on the scanning bed for 20 minutes;

Exclusion Criteria:

1. Known allergic history to 68Ga FAPI or its excipients;
2. Patients who can not tolerate intravenous drug administration (such as needle fainting and blood fainting history);
3. Those who are not suitable for or unable to complete imaging tests such as PET due to special reasons, including claustrophobia and radiophobia;
4. pregnant and lactating women;
5. Workers who are exposed to radiation for a long period of time;
6. Serious diseases of the heart, kidney, lung, blood vessel, nervous system, mental system, immune deficiency diseases and hepatitis/cirrhosis;
7. Participating in other interventional clinical trials within 1 month before screening;
8. Patients undergoing chemotherapy, immunotherapy or molecular targeted therapy due to other cancers;
9. There are other circumstances that the researcher thinks are not suitable for participating in this study;

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Chinese people
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2023-11-22 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Sensitivity | Up to 24 months
  Sensitivity of 68Ga-FAPI PET/CT Imaging for the detection of Myelofibrosis.
Specificity | Up to 24 months
  Specificity of 68Ga-FAPI PET/CT Imaging for the detection of Myelofibrosis.
Positive prediction rate | Up to 24 months
  Positive prediction rate of 68Ga-FAPI PET/CT Imaging for the detection of Myelofibrosis.
Negative prediction rate | Up to 24 months
  Negative prediction rate of 68Ga-FAPI PET/CT Imaging for the detection of Myelofibrosis.

CONTACTS AND LOCATIONS:
Overall Officials: Bing Xu, Principal Investigator — The First Aiffiliated hosptical of xiamen University
Locations (1):
- Bing Xu, Xiamen, Fujian, China

IPD SHARING:
Plan to Share IPD: No